CLINICAL TRIAL: NCT00484757
Title: Effect of Intranasal Administration of Orexine A on IL-6-System, Sleep-Wake-Regulation and Neurocognition
Acronym: NARKOREX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zentrum für Integrative Psychiatrie (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Narkorex; DFG-SFB654/C5-Narkorex
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; Orexines; sleep; cognition; cytokines
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Orexine A

SUMMARY:
15 patients with narcolepsy and 15 healthy controls will be included in the study. According to a randomized, double-blind protocol they will receive intranasally at night first Orexine A and approximately two weeks later placebo or vice versa. Thereafter sleep will be recorded, the cytokine-system and neurocognition characterized.

ELIGIBILITY:
Inclusion Criteria:

* Narcolepsy
* Age >18
* Informed consent
* GERMAN fluently spoken

Exclusion Criteria:

* Additional severe psychiatric or somatic disorders
* Pregnancy or nursing
* Anemia (Hb<10g/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-06; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Effect of orexine A on sleep, neurocognition and immune-system

CONTACTS AND LOCATIONS:
Overall Officials: Dunja Hinze-Selch, MD, Principal Investigator — Zentrum für Integrative Psychiatrie
Locations (1):
- Zentrum für Integrative Psychiatrie, Kiel, Germany